CLINICAL TRIAL: NCT04096872
Title: Clinical Application of Laparo-endoscopic Single-site Surgery and Natural Orifice Transluminal Endoscopic in Gynecology- the Chinese National Registry
Brief Title: Clinical Application of Laparo-endoscopic Single-site Surgery and Natural Orifice Transluminal Endoscopic in Gynecology
Acronym: GLESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese Medical Doctor Association (Other); Chinese Obstetricians and Gynecologists Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: GLESS-NOTES.CN
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Cervical Cancer, Endometrial Cancer，Endometrial Lesion & Adnexal Lesion，Ectopic Pregnancy & Infertility，Pelvic Obstructive Disorder & Genital Tract Deformity
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The GLESS registry is a prospective multi-center observational registry. Data from the time of patient admission, operation, discharge, and follow-up will be collected for this registry. Eight gynecological conditions included were: cervical cancer, endometrial cancer, endometrial lesion, adnexal lesion, ectopic pregnancy, infertility, pelvic obstructive disorder, and genital tract deformity.

DETAILED DESCRIPTION:
Founding of the group. In June 2016 with the support of the Chinese Medical Doctor's Association and Chinese OBGYN Association, the not-for-profit GLESS (including Notes) Working Group was founded. The national Working Group is tasked with creating and maintaining the Prospective GLESS data registry, standardizing LESS surgeon training, creating best practices and guidelines. The Working Group aims to extend to all 35 provinces in Mainland China covering over 200 hospitals nationwide.

The GLESS Working Group published an expert consensus in 2017 on the indications and contraindications of the surgery. The GLESS registry is a prospective observational case-only database. Literature has cases, outcomes are positive and promising, but there lacks a systematic and large scale multi-center registry to provide data driven evidence for best practices.

The goal for the group (evidence level- can we achieve level 1, Canada task force). Research, share experiences to identify indications, standard surgical practices, understand outcomes/observations. Provide empirical evidence for GLESS and Notes surgical indications and complications. Provide empirical evidence for advancing procedures, expanding surgical indications (e.g. can GLESS be performed on cervical cancer?), what is the reliability, standard procedures for training Create best practices for 1)Identifying suitable clinical indications- expanding 2)surgical techniques (entry, port placement, trochar, retraction, suture, ligation) & selecting surgical instrumentation3)Identifying, minimizing, and handling complications.

4)Carrying out optimal perioperative and postoperative care 5)Creating a safe and comfortable experience in terms of cosmesis, pain, and overall experience 6)Understand how various techniques can impact short/mid/long term for patients Outcomes will include a National effort to coordinate followup to create the largest/most reliable data set for understanding prognostic outcomes related to GLESS. With accumulated data/big data techniques develop comprehensive short term and long term scoring systems for colleagues and patients around the world. Create standard nomenclature for easier collaboration and communication between gynecologists Note on NOTES? Why we include it here. Yes, notes is a natural progression from LESS. With the orifice being the vagina. We believe understanding the risks/rewards of such a procedure can make the transition from an umbilical to vaginal entry point easy.

ELIGIBILITY:
Inclusion Criteria:

- Adults over 18 years of age, that have the conditions eligibility with severity meeting within the surgical indications of the 2017 Chinese expert consensus on GLESS. Eligibility will be confirmed by the gynecological surgeon who are treating at each location. Patients are recruited after admission and prior to the operation.

Exclusion Criteria:

1. Acute infection stage, preoperative deep venous thrombosis or hypercoagulability, fasting blood sugar > 11.1 mmol/L, blood pressure > 160/100 mmHg, liver and kidney dysfunction, mental illness and other surgical contraindications;
2. Refuse to sign informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — GLESS- A National Gynecological laparoendoscopic single site surgery registry
Study Population: Types of conditions included in the GLESS registry. Malignancies:Cervical cancer, Endometrial cancer Benign lesion：Endometrial lesion & Adnexal lesion Reproductive conditions：Ectopic pregnancy & infertility Structural abnormalities/lesions：Pelvic obstructive disorder & Genital tract deformity
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Completion time | One time (intraoperative)
Success rate | One time (intraoperative)
Recurrence rate | 36 months
Conversion rate | One time (intraoperative)

CONTACTS AND LOCATIONS:
Locations (1):
- Gless-Notes, Beijing, Beijing Municipality, China